CLINICAL TRIAL: NCT01841320
Title: Seek, Test, Treat Strategies for Vietnamese Drug Users: A Randomized Controlled Trial
Acronym: VISTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Hanoi Center for HIV/AIDS Prevention and Control (Unknown)
Responsible Party: Principal Investigator, Vu Minh Quan, Assistant Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: R01DA030776 (NIH)
Record Dates: First submitted 2013-04-24; First posted 2013-04-26 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: HIV; Addiction
MeSH Terms: conditions — Behavior, Addictive | interventions — Ambulatory Care Facilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Participants who are assigned to intervention arm will receive ART and methadone maintenance at an integrated methadone and antiretroviral therapy (iMART) clinic and ART adherence support through the use of mobile phone technologies.
  Interventions: Other: Integrated methadone and antiretroviral therapy (iMART) clinic
- Standard of Care (No Intervention): Participants will be referred to standard HIV outpatient clinics and methadone maintenance clinics.

INTERVENTIONS:
Other: Integrated methadone and antiretroviral therapy (iMART) clinic
  Other Names: ART access support; ART adherence support through mobile phone technologies
  Arms: Intervention

SUMMARY:
This research examines the effectiveness of an intervention that employs seek, test, and treat strategies for Vietnamese injection drug users (IDU) and their network members, by ensuring that high risk individuals are sought for HIV testing and promptly referred to and maintained on antiretroviral therapy (ART). HIV prevention interventions are provided to IDUs who test HIV-negative, as well as those who test HIV-positive. HIV-positive IDUs will be referred to HIV care through a two-arm randomized controlled trial to compare the effects of different levels of engagement in care on ART uptake, ART adherence, and treatment outcome.

DETAILED DESCRIPTION:
Opioid injection and HIV infection are major public health problems in Vietnam. Injection drug users (IDUs) have a high burden of HIV infection (20% HIV prevalence, nationally; 6% mortality per year) and the high rate of HIV transmission continues (HIV incidence, 5% per year). The investigators propose an intervention that employs the seek, test, and treat strategies for the IDU population and their network members, by ensuring that high risk individuals are sought for HIV testing, promptly referred to and maintained on ART, while HIV prevention interventions provided to the many who test HIV-negative, as well as those who test HIV-positive. The intervention will seek and test IDUs and their network members in the community, particularly those who are recently released from drug treatment centers. HIV-positive IDUs will be referred to HIV care through a two arm randomized controlled trial to compare the effects of different levels of engagement in care on ART uptake, antiretroviral adherence, and treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Recently released from drug treatment centers;
3. Positive HIV serology;
4. Male;
5. Meet criteria for ART initiation according to Vietnam's national guidelines;
6. Provide informed consent for the study; and
7. Reside in study area and do not plan to move away in the next 18 months.

Exclusion Criteria:

1. Currently on ART;
2. Co-enrollment in other HIV interventional research study;
3. Unwilling to provide locator information.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2011-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Time from randomization to the initiation of antiretroviral therapy (ART) | At month 3

SECONDARY OUTCOMES:
CD4+ counts | At months 6, 12, and 18
HIV-1 RNA levels | At months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Quan M Vu, M.D, Principal Investigator — Johns Hopkins University
Locations (1):
- Tu Liem Medical Center, Hanoi, Vietnam